CLINICAL TRIAL: NCT01499225
Title: A Double-blind, Randomized, Parallel, Placebo-active Controlled, Multi-center Phase II Clinical Trial to Investigate the Efficacy and Safety of YH14642 Following 12-week Oral Administration in Patients With Chronic Periodontal Disease
Brief Title: A Clinical Trial of YH14642 in Patients With Chronic Periodontal Disease
Acronym: YH14642
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH14642-201
Record Dates: First submitted 2011-12-13; First posted 2011-12-26 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Capsules

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- YH14642 A-I (Experimental)
  Interventions: Drug: YH14642 500mg Tab
- YH14642 A-II (Experimental)
  Interventions: Drug: YH14642 500mg Tab
- YH14642 A-III (Experimental)
  Interventions: Drug: YH14642 500mg Tab
- Active Comparator B (Active Comparator)
  Interventions: Drug: INSADOL[Zea mays L. extract] 35mg Tab
- Active Comparator C (Active Comparator)
  Interventions: Drug: DENTISTA[Doxycycline hyclate] 20mg Cap
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH14642 500mg Tab — YH14642 500mg per day(once a day)
  Arms: YH14642 A-I
Drug: YH14642 500mg Tab — YH14642 1000mg per day(twice a day)
  Arms: YH14642 A-II
Drug: YH14642 500mg Tab — YH14642 2000mg per day(three times a day)
  Arms: YH14642 A-III
Drug: INSADOL[Zea mays L. extract] 35mg Tab — [Initiation dose : 4weeks after administraion] INSADOL[Zea mays L. extract] 210mg TAB per day
  [Maintain dose : Between 4weeks and 8weeks after administraion] INSADOL[Zea mays L. extract] 105mg TAB per day
  [Maintain dose : Between 8weeks and 12weeks after administraion] INSADOL[Zea mays L. extract] 105mg TAB per day
  Arms: Active Comparator B
Drug: DENTISTA[Doxycycline hyclate] 20mg Cap — DENTISTA[Doxycycline hyclate] Cap 40mg per day
  Arms: Active Comparator C
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and the safety of YH14642 in Korea patients with chronic periodontitis, in order to investigate the recommended therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 20 years of age or older
* Have at least 18 natural teeth
* Four or more clinical attachment level(CAL) ≥ 3mm
* Four or more periodontal pockets with a probing depth (PD) ≥ 4mm
* Have Bleeding on probing
* Provide informed consent and willingness to cooperate with the study protocol

Exclusion Criteria:

* Forbidden History of Panax Notoginseng and Rehmanniae Radix Preparata
* Hypersensitivity of Doxycycline
* Hypersensitivity of Zea mays L. extract
* Critical diseases such as HIV previous three years
* Patients with mental retardation and dementia
* Systemic diseases such as diabetes and hypertension
* Patients who take Anticoagulants or Antiplatelet Agents
* Patients who have malignant tumor
* Smoker
* Continually use for 2weeks of phenytoin, calcium channel blocker, cyclosporin, coumarin, nonsteroidal anti-inflammatory drugs and aspirin use in the previous one month
* Patients who need malignant tumor
* Patients who received periodontal treatment within the last 6 months
* Pregnant or lactating females

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in probing pocket depth (PD) | baseline, 4weeks, 8weeks and 12weeks

SECONDARY OUTCOMES:
Change in Clinical attachment level (CAL) | baseline, 4weeks, 8weeks and 12weeks
Change in Bleeding on probing(BOP) | baseline, 4weeks, 8weeks and 12weeks
change in Gingival index(GI) | baseline, 4weeks, 8weeks and 12weeks
Change in Plaque index (PI) | baseline, 4weeks, 8weeks and 12weeks
Change in Gingival recession(GR) | baseline, 4weeks, 8weeks and 12weeks
[Exploratory Outcome Measure] Change in Alveolar bone height(ABH) | baseline and 12weeks
[Exploratory Outcome Measure] Change in Alveolar bone density(ABD) | baseline and 12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Dental Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289